CLINICAL TRIAL: NCT02872129
Title: 12-years Follow-up on 166 Female Patients With Fibromyalgia or Chronic Widespread Pain
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: GAU1-U
Record Dates: First submitted 2016-06-30; First posted 2016-08-19 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Fibromyalgia; Chronic Widespread Pain
Keywords: Fibromyalgia; chronic widespread pain; follow-up; pain; fatigue; symptoms; workability; physical function
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Pain; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 166 women with FM/CWP: 166 women with Fibromyalgia (FM) or Chronic Widespread Pain (CWP) that participated in an Randomised Controlled Trial called GAU in western Sweden 2004-2005.

SUMMARY:
A 12-year follow-up of 166 women with fibromyalgia (FM) or chronic widespread pain (CWP) in western Sweden.

The 166 women participated in a Randomised Controlled Trial called GAU in 2004-2005, aiming to investigate the effect of pool exercise and patient education.

The primary aim of the present study is to examine the change of symptoms after 11-12 years in 166 women with FM or CWP and also investigate predictors of change of symptoms and work ability.

The 166 women will be asked to participate in the present follow-up study. The follow-up examination comprises a standardised interview of symptoms and demographic variables, a battery of self-administered questionnaires and tests of physical function.

DETAILED DESCRIPTION:
A 12-year follow-up of 166 women with fibromyalgia (FM) or chronic widespread pain (CWP).

The 166 women participated in a Randomised Controlled Trial called GAU 2004-2005 in three cities in western Sweden; Göteborg, Alingsås and Uddevalla. The RCT aimed to investigate the effect of pool exercise and patient education.

The primary aim of the present study is to examine the change of symptoms after 11-12 years in 166 women with FM or CWP and also investigate predictors of change of symptoms and work ability.

The 166 women will be contacted by mail and telephone, and asked to participate in the present follow-up study.

The follow-up examination comprises a standardised interview of symptoms and demographic variables, a battery of self-administered questionnaires and tests of physical function.

ELIGIBILITY:
Inclusion Criteria of the present study GAU-U:

* All 166 patients who participated in the study GAU in 2004/2005. (The inclusion criteria of GAU was women with FM or CWP, 18-60 years old. Patients with widespread pain; pain in the right and left side of the body, above and below the waist, as well as axial pain, for at least three months were classified as chronic widespread pain (CWP). Patients who fulfilled the criteria for CWP and who also had pain at palpation of at least 11 of 18 pre-defined tender points were classified as fibromyalgia (FM).

Exclusion criteria for GAU was serious physical or psychological disease)

Exclusion Criteria of the present study GAU-U:

* Patients who has developed serious physical or psychological disease since participating in the GAU 2004/2005

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 166 women who 2004/2005 participated in the study GAU.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
pain intensity | 2016 (to be compared with previous examination performed in 2004/2005)
  pain intensity assessed with the Fibromyalgia Impact questionnaire subscale for pain
distribution of pain | 2016 (to be compared with previous examination performed in 2004/2005)
  Distribution of pain

SECONDARY OUTCOMES:
Fatigue | 2016 (to be compared with previous examination performed in 2004/2005)
  fatigue assessed with the Multidimensional fatigue inventory (MFI-20)
Fatigue | 2016 (to be compared with previous examination performed in 2004/2005)
  fatigue assessed with the Fibromyalgia Impact Questionnaire subscale for global fatigue
workability | 2016 (to be compared with previous examination performed in 2004/2005)
  workability assessed as percentage of full time in work
Walking capacity | 2016 (to be compared with previous examination performed in 2004/2005)
  Walking capacity assessed with 6 min walk test
Physical function in lower limbs | 2016 (to be compared with previous examination performed in 2004/2005)
  physical function in lower limbs assessed with chair-test
Hand grip force | 2016 (to be compared with previous examination performed in 2004/2005)
  Hand grip force assessed with the Grippit
Physical activity | 2016 (to be compared with previous examination performed in 2004/2005)
  physical activity in leisure time assessed with the Leisure Time Physical Activity Instrument
Depression and anxiety | 2016 (to be compared with previous examination performed in 2004/2005)
  depression and anxiety assessed with the Hospital Anxiety and Depression Scale
Health related quality of life | 2016 (to be compared with previous examination performed in 2004/2005)
  Health related quality of life assessed with the Short-Form 36

OTHER OUTCOMES:
sleep | 2016 (to be compared with previous examination performed in 2004/2005)
  quantity and quality of sleep
alcohol consumption | 2016 (to be compared with previous examination performed in 2004/2005)
  alcohol consumption assessed with the Balogh questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bergenheim, PhD, Study Director — University of Gothenburg, Sahlgrenska Academy, Institution of Neuroscience and Physiology - Section of Health and Rehabilitation, Physiotherapy, Göteborg, Sweden
Locations (3):
- Sweden (3):
  - Närhälsan, Region Västra Götaland, Alingsås
  - Närhälsan, Region Västra Götaland, Gothenburg
  - Närhälsan, Region Västra Götaland, Uddevalla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergenheim A, Juhlin S, Nordeman L, Joelsson M, Mannerkorpi K. Stress levels predict substantial improvement in pain intensity after 10 to 12 years in women with fibromyalgia and chronic widespread pain: a cohort study. BMC Rheumatol. 2019 Jun 24;3:5. doi: 10.1186/s41927-019-0072-9. eCollection 2019. PMID 31286111